CLINICAL TRIAL: NCT02232308
Title: Modulation of Heme Oxygenase 1 by Nizatidine and Lisinopril in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Adil Bharucha (Other)
Collaborators: National Center for Research Resources (NCRR) (NIH); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor-Investigator, Adil Bharucha, Professor of Medicine, Mayo Clinic
Organization: Mayo Clinic (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 14-004137; UL1RR024150 (NIH); P01DK068055 (NIH)
Record Dates: First submitted 2014-06-23; First posted 2014-09-05 (Estimated); Last update posted 2015-04-30 (Estimated); Status verified 2015-04

CONDITIONS: Gastroparesis
MeSH Terms: conditions — Gastroparesis | interventions — Nizatidine; Lisinopril

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Nizatidine (Experimental): Nizatidine (150 mg) will be administered once daily for the first 3 days, then twice daily for days 4-9, and once on day 10.
  Interventions: Drug: Nizatidine
- Lisinopril (Experimental): Lisinopril (10 mg) will be administered once daily for the first 3 days, then twice daily for days 4-9, and once on day 10.
  Interventions: Drug: Lisinopril
- Nizatidine plus Lisinopril (Experimental): Nizatidine (150 mg) and Lisinopril (10 mg) will be administered once daily for the first 3 days, then twice daily for days 4-9, and once on day 10.
  Interventions: Drug: Nizatidine; Drug: Lisinopril
- Placebo (Placebo Comparator): Placebo capsules to match active drug will be administered once daily for the first 3 days, then twice daily for days 4-9, and once on day 10.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Nizatidine — Nizatidine (150 mg) will be administered once daily for the first 3 days, then twice daily for days 4-9, and once on day 10.
  Other Names: Axid
  Arms: Nizatidine; Nizatidine plus Lisinopril
Drug: Lisinopril — Lisinopril (10 mg) will be administered once daily for the first 3 days, then twice daily for days 4-9, and once on day 10.
  Other Names: Zestril; Prinivil
  Arms: Lisinopril; Nizatidine plus Lisinopril
Drug: Placebo — Placebo capsules to match active drug will be administered once daily for the first 3 days, then twice daily for days 4-9, and once on day 10.
  Arms: Placebo

SUMMARY:
To assess if oral nizatidine or lisinopril alone and in combination will increase heme oxygenase 1 (HO-1) protein concentration and activity compared to placebo in healthy subjects.

DETAILED DESCRIPTION:
Current therapeutic options for gastroparesis are limited to dietary modifications and pharmacological (i.e., prokinetic and symptomatic) agents. Exciting and novel preliminary data from our programs demonstrate that (i) reduced expression of heme oxygenase 1 (HO-1) is responsible for loss of interstitial cells of Cajal and delayed gastric emptying in non-obese diabetic (NOD) mice, (ii) upregulation of (HO-1) reverses delayed gastric emptying in this model, perhaps by generating carbon monoxide (CO), which has anti-apoptotic and cytoprotective actions, and may relax smooth muscle, and (iii) hemin upregulates HO-1 in humans. However, hemin is exorbitant and can only be administered intravenously. A large throughput screening assay uncovered that the histamine H2 receptor antagonist nizatidine and the ACE inhibitor lisinopril upregulate HO-1 in Human Embryonic Kidney (HEK) cells. Hence, this double-blind placebo-controlled study will randomly assign 24 healthy subjects to one of 4 arms, and HO-1 protein activity and concentration will be assessed.

ELIGIBILITY:
Inclusion criteria:

* Healthy subjects without clinical evidence of significant cardiovascular, gastrointestinal, hematological, neurological, psychiatric or other disease that may interfere with the objectives of the study and/or pose safety concerns
* Normal serum potassium and estimated glomerular filtration rate (eGFR) > 60 ml/minute
* Baseline systolic BP ≥ 110 mmHg
* No known hypersensitivity to lisinopril or nizatidine
* Able to provide written informed consent before participating in the study
* Able to communicate adequately with the investigator and to comply with the requirements for the entire study.

Exclusion criteria:

* Pregnant
* Breast feeding
* Current smoker
* Symptoms of functional GI disorder as assessed by a validated questionnaire
* Previous history of peptic ulcer disease.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2014-07; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Change in plasma heme oxygenase 1 (HO-1) protein concentration | Day 3, Day 10
  Heme oxygenase (HO-1) degrades heme and protects against oxidative stress. HO-1 concentration was measured by a blood test; the units are ng/ml.
Change in Monocyte HO-1 activity | Day 3, Day 10
  Heme oxygenase (HO-1) degrades heme and protects against oxidative stress. When HO-1 is induced, more heme is removed, and end products of heme metabolism (i.e., carbon monoxide, iron, and bilirubin) are generated. HO-1 activity was measured by a blood test, the units are pmol bilirubin/mg/h.

CONTACTS AND LOCATIONS:
Overall Officials: Adil Bharucha, MBBS, MD, Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Mayo Clinic, Rochester, Minnesota